CLINICAL TRIAL: NCT00628654
Title: Clinical Protocol to Evaluate Glycans Analysis As a Diagnostic Test for Ovarian Cancer
Brief Title: Glycan Analysis in Diagnosing Cancer in Women With Ovarian Epithelial Cancer and in Healthy Female Participants
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 251975; CDR0000583063 (Other: UC Davis IRB); UCD-183 (Other: University of California Davis); UCD-200513707 (Other: University of California Davis); P30CA093373 (NIH)
Record Dates: First submitted 2008-03-04; First posted 2008-03-05 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer
Keywords: ovarian germ cell tumor; ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Volunteers: Serum samples will be obtained from volunteers, but no tissue specimens. Volunteers will complete a questionnaire.
- Patients with cancer: Ascites from patients with ovarian, peritoneal, and fallopian tube cancers for basic science studies

SUMMARY:
RATIONALE: New diagnostic procedures, such as glycan analysis, may be effective in finding ovarian epithelial cancer.

PURPOSE: This clinical trial is studying how well glycan analysis works in diagnosing cancer in women with ovarian epithelial cancer and in healthy female participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the accuracy of glycan analysis to distinguish between normal healthy control female subjects and those with ovarian epithelial cancer.

Secondary

* Compare the new assay to the standard CA 125 for diagnostic accuracy.

OUTLINE:

* Ovarian cancer patients: Blood samples are obtained periodically for up to 2 years. Patients undergoing surgery have blood samples drawn before and after surgery. Medical charts are reviewed periodically for up to 3 years.
* Healthy volunteers: One blood sample is obtained. Volunteers also complete a 1-page questionnaire.

PROJECTED ACCRUAL: A total of 300 healthy female participants and 400 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand consent document for participation in the study
* Not pregnant
* Negative pregnancy test

Participants must meet 1 of the following criteria:

* Patients scheduled for ovarian surgery for an ovarian mass
* Healthy female volunteers with no active cancer or history of cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: volunteers and patients with ovarian, peritoneal, and fallopian tube cancers
Sampling Method: Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2005-10; Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of glycan analysis | one time for healthy volunteers; up to 2 years for patients with cancer
  For healthy controls, a single sample will be obtained. For patients scheduled for surgery, two samples will be obtained: one preoperatively and one postoperatively. Ovarian cancer patients who agree to participate in the longitudinal study will have follow-up serum samples drawn periodically during chemotherapy treatments and then during surveillance visits, to correspond with routine blood testing for CA 125. They will be asked to participate for 2 years, with a maximum of 8 blood draws per year (to be coordinated with other venipunctures, if possible).

SECONDARY OUTCOMES:
Comparison of the new assay to the standard CA 125 assay | one time for healthy volunteers; up to 2 years for patients with cancer
  For healthy controls, a single sample will be obtained. For patients scheduled for surgery, two samples will be obtained: one preoperatively and one postoperatively. Ovarian cancer patients who agree to participate in the longitudinal study will have follow-up serum samples drawn periodically during chemotherapy treatments and then during surveillance visits, to correspond with routine blood testing for CA 125. They will be asked to participate for 2 years, with a maximum of 8 blood draws per year (to be coordinated with other venipunctures, if possible).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Leiserowitz, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States